CLINICAL TRIAL: NCT04745533
Title: Diagnostic Efficacy of the SARS-CoV2 Antigen Detection Test for the COVID-19 Contact Study
Brief Title: COVID-19 Contact Study by Antigen Detection Test
Acronym: DETAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Juan Fernando Masa Jiménez (Other)
Responsible Party: Sponsor-Investigator, Juan Fernando Masa Jiménez, Principal investigator, University of Extremadura
Organization: University of Extremadura (Other)
Other Study IDs: 12/2020
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV Infection
Keywords: Antigen detection tests; Diagnostic efficacy; Contact study; Asymptomatic contacts
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV2 contacts: Subjects considered close contacts of COVID-19 patients according to the definition of the Ministry of Health in the health area of Cáceres.
  Interventions: Diagnostic Test: Antigen detection test

INTERVENTIONS:
Diagnostic Test: Antigen detection test — To compare the results of the antigen detection test against the polymerase chain reaction in the study of contacts of COVID-19 patients during quarantine.

SUMMARY:
Stopping the SARS-CoV2 spread is essential to control the pandemic cause by this virus.

A great effort is being made to carry out surveillance, case detection and contact control protocols in order to detect and isolate those contagious subjects.

Since both symptomatic and asymptomatic subjects can be contagious, a surveillance system based on the presence of symptoms is not enough, requiring to perform diagnostic tests in a large number of subjects, such as asymptomatic contacts or high-prevalence populations, and repeatedly. Moreover, the speed in obtaining results is crucial in order not to delay the isolations of positive subjects.

The polymerase chain reaction (PCR) is an expensive test which requires specialized equipment and personnel with a delay in results of 24-48 hours. In addition, its high sensitivity can mean that subjects without infective capacity have a positive result.

In contrast, antigen detection tests (ADTs) are cheap and easy to perform, having a result in few minutes. They have shown high sensitivity and specificity in symptomatic subjects, specially in the first week of symptoms when the viral load is high. This could be very useful for the study of asymptomatic contacts to detect those with potential contagiousness quick, easily and cheaply. However, there is no evidence to support the use of ADTs in this group of subjects.

For this reason, the investigators propose to carry out a study to compare the diagnostic efficacy of ADTs versus PCR in the group of subjects considered to be close contacts of SARS-Cov2 positive patients in the health area of Cáceres.

ELIGIBILITY:
Inclusion Criteria:

* Subjects considered close contacts of COVID-19 patients according to the definition of the Ministry of Health of Spain at the time of inclusion.

Exclusion Criteria:

* Subjects who do not obtain their informed consent for the study.
* Symptomatic subject at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects considered close contacts of COVID-19 patients according to the definition of the Ministry of Health of Spain in the health area of Cáceres
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the antigen detection test used in the study of contacts of COVID-19 patients. | 2 days
  The investigators will analyze the probability of a positive antigen detection test result in a COVID-19 patient contact with a positive polymerase chain reaction test.
Specificity of the antigen detection test used in the study of contacts of COVID-19 patients. | 2 days
  The investigators will analyze the probability of a negative antigen detection test result in a COVID-19 patient contact with a negative polymerase chain reaction test.

SECONDARY OUTCOMES:
Positive predictive value of the antigen detection test used in the study of contacts of COVID-19 patients. | 2 days
  The investigators will analyze the probability that a subject considered COVID-19 patient contact with a positive antigen detection test result has a positive polymerase chain reaction test.
Negative predictive value of the antigen detection test used in the study of contacts of COVID-19 patients. | 2 days
  The investigators will analyze the probability that a subject considered COVID-19 patient contact with a negative antigen detection test result has a negative polymerase chain reaction test.
Positive likelihood ratio of the antigen detection test used in the study of contacts of COVID-19 patients. | 2 days
  The investigators will analyze how much the probability of having a positive polymerase chain reaction test increases when a subject considered a COVID-19 patient contact has a positive antigen detection test.
Negative likelihood ratio of the antigen detection test used in the study of contacts of COVID-19 patients. | 2 days
  The investigators will analyze how much the probability of having a positive polymerase chain reaction test decreases when a subject considered a COVID-19 patient contact has a negative antigen detection test.
Change in the pretest probability when the antigen detection test result is positive in a COVID-19 patient contact. | 2 days
  The investigators will analyze the change that occurs in the probability that a subject considered a COVID-19 contact has a positive polymerase chain reaction test before and after performing an antigen detection test with a positive result
Change in the pretest probability when the antigen detection test result is negative in a COVID-19 patient contact. | 2 days
  The investigators will analyze the change that occurs in the probability that a subject considered a COVID-19 contact has a positive polymerase chain reaction test before and after performing an antigen detection test with a negative result
Cut-off point of the cycle threshold of the polymerase chain reaction test that discriminates infectivity. | 2 weeks
  The investigators will analyze the cut-off point of polymerase chain reaction test (PCR) cycle threshold that maximizes discrimination of patients with at least one close contact with positive PCR (infectivity in the first circle of contacts).
Risk of SARS-CoV2 infection in close contacts of COVID-19 patients with a positive polymerase chain reaction test depending on whether the antigen detection test is positive or negative. | 2 weeks
  The investigators will compare the number of infected subjects by COVID-19 patient contacts with a positive polymerase chain reaction test, depending on whether the antigen detection test is positive or negative
To predict a positive result of the polymerase chain reaction test based on the appearance of symptoms during quarantine | 10 days
  Researchers will analyze the appearance of symptoms during quarantine in the contacts of COVID-19 patients and whether or not they have a positive polymerase chain reaction test.
The percentage of COVID-19 patient contacts with symptoms during the quarantine. | 10 days
  The investigators analyze the percentage of contacts of COVID-19 patients who develop symptoms during the quarantine.

IPD SHARING:
Plan to Share IPD: Yes
Additional related documents such as study protocol, statistical analysis plan and informed consent form will be available upon request from the project principal investigator.
  (Dr. Juan Fernando Masa Jiménez). De-identified patients´data can be requested by researchers for use in independent scientific research and will provided following review and approval of the research proposal (including statistical analysis plan) and completion of a data sharing agreement with the Project Publications Committee. Investigator Data requests can be made anytime from 1 to 2 years after the publication of this trial. Requests should be sent to the corresponding author (Dr. Juan Fernando Masa Jiménez- fmasa@separ.es)